CLINICAL TRIAL: NCT06440798
Title: Examining the Effects of Mental Health Content on Help-Seeking and Self-Diagnosing Behavior: Cross-sectional Survey Study
Brief Title: Mental Health Content and Mental Health Outcomes
Status: Recruiting | Type: Observational
Sponsor: Yale-NUS College (Other)
Responsible Party: Sponsor
Other Study IDs: NUS-IRB-2023-864
Record Dates: First submitted 2024-05-27; First posted 2024-06-04 (Actual); Last update posted 2024-06-04 (Actual); Status verified 2024-06

CONDITIONS: Help-Seeking Behavior; Psych; Depression; Anxiety; Stress
Keywords: Mental Health Content
MeSH Terms: conditions — Help-Seeking Behavior; Depression; Anxiety Disorders

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The study will aim to explore the relationship between mental health content on social media and health behavior, addressing a gap in empirical research. Using the Theory of Planned Behavior, a survey with over 600 participants will examine associations between exposure to mental health content and behaviors like help-seeking and self-diagnosis.

DETAILED DESCRIPTION:
Background: Mental health content has recently surged in popularity across social media. However, current empirical research lacks a comprehensive understanding of the relationship between mental health content and health behaviour.

Objective: This study will aim to address this gap by examining different types of mental health content and their relationship to behavior. Specifically, it will explore whether exposure to mental health content will be associated with either positive behaviors, like help-seeking, or maladaptive ones, such as self-diagnosing.

Methods: Utilizing the Theory of Planned Behavior, a cross-sectional epidemiological survey will be conducted with over 600 participants to answer the research questions. Baseline measures will include participants' exposure to various types of mental health content, and mental well-being (depression, anxiety, and scores from the DASS-21). The outcome measures of interest will be help-seeking attitude (IASMHS) and self-diagnosing (SELF-I) behavior.

ELIGIBILITY:
Inclusion Criteria:

* Enrollment is restricted to healthy adults between 21-34 (or 18-34 for university students)
* Use at least one social media platform (e.g., Facebook, Instagram, LinkedIn, X)
* Participants need to be able to read and understand English.
* Participants must also have lived in Singapore for at least 2 years.

Exclusion Criteria:

* Anyone who does not feel comfortable answering questions related to mental health and exposure to mental health-related content online.

Ages: 18 Years to 34 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Recruiting a representative sample of around 600 people through the National University of Singapore (NUS) and the general public in Singapore through physical posters or online platforms (e.g., the university's Work Scheme website, and research groups on Telegram).
Sampling Method: Non-Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2024-01-01 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Help-Seeking Behaviors | Through study completion, an average of 1 year
  Inventory of Attitudes toward Seeking Mental Health Services (IASMHS). Items were on a 5-point Likert scale ranging from 0 ("Somewhat Disagree") to 4 ("Agree").
Self-Diagnosing Behaviors for Mental Health | Through study completion, an average of 1 year
  Self-identification as having a Mental Illness (SELF-I) scale. Items were on 5-point Likert scale ranging from 1 (Not true at all) to 5 (Completely True)

CONTACTS AND LOCATIONS:
Overall Officials: Sundarimaa Erdembileg, Principal Investigator — Yale-NUS College
Locations (1):
- Yale-NUS, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No
Given the sensitivity of mental health disclosures and the age of the population, no individual participant data will be shared as agreed upon with the IRB. Results will be published by the investigators in academic journals. Sharing of generated study data can be made available upon request by writing to the investigator(s).